CLINICAL TRIAL: NCT07263412
Title: A Multicenter Prospective Cohort Study to Identify Risk Factors and Develop a Diagnostic Prediction Model for Gestational Diabetes Mellitus, and to Evaluate the Effectiveness of Multidisciplinary Precision Health Interventions (GLOW Plan)
Brief Title: Gestational Lifestyle & Outcomes Wellness
Status: Recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: GLOW-GDM-COHORT-2024
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-10

CONDITIONS: GDM
MeSH Terms: interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- CGM group
  Interventions: Device: cgm
- SMBG group
  Interventions: Behavioral: Behavioral Self-Monitoring of Blood Glucose
- Control group
  Interventions: Other: Control

INTERVENTIONS:
Device: cgm — Participants will wear a continuous glucose monitoring device to continuously record glucose levels throughout the study period, in addition to receiving standard prenatal care.
  Groups: CGM group
Behavioral: Behavioral Self-Monitoring of Blood Glucose — Participants will perform regular self-monitoring of blood glucose using a finger-prick glucose meter, along with standard prenatal care.
  Groups: SMBG group
Other: Control — Participants will receive standard prenatal care without additional glucose monitoring interventions
  Groups: Control group

SUMMARY:
A Multicenter Prospective Cohort Study to Identify Risk Factors and Develop a Diagnostic Prediction Model for Gestational Diabetes Mellitus, and to Evaluate the Effectiveness of Multidisciplinary Precision Health Interventions (GLOW Plan)

ELIGIBILITY:
Inclusion Criteria: All must be met

1. Aged 18-40 years;
2. Pre-pregnancy BMI: 18.5 kg/m² < BMI < 28 kg/m²;
3. Able to read, understand and sign the informed consent form;
4. Receive prenatal care and deliver in the study hospital.

Exclusion Criteria: Any one met leads to exclusion

1. Twin or multiple pregnancies;
2. Pre-gestational diabetes mellitus (PGDM), including new-onset diabetes during pregnancy;
3. Poorly controlled pre-pregnancy chronic hypertension (BP ≥140/90 mmHg);
4. Complicated with severe liver/kidney diseases;
5. Current/recent use of drugs affecting glucose metabolism;
6. Mental illness or severe psychological disorders;
7. Complicated with severe infection;
8. Poor compliance or refusal to use CGM/SMBG.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: A total of 1,000 pregnant women with antenatal care registration in the study hospital are enrolled, including 500 Gestational Diabetes Mellitus (GDM) cases (diagnosed via 75g OGTT at 24-28 weeks of gestation with ≥1 abnormal blood glucose value) and 500 normal controls.
  All participants meet: aged 18-40 years, pre-pregnancy BMI 18.5-28 kg/m², ability to sign informed consent, and prenatal care/delivery in the hospital. Those with multiple pregnancies, pre-gestational diabetes, poorly controlled hypertension, severe organ diseases, or poor compliance are excluded. Participants and their offspring complete perinatal and 2-year postnatal follow-ups.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Improvement Rate of Glucose Metabolism During the Perinatal Period | From participant enrollment (23-24+6 weeks of gestation) to 6 weeks postpartum.

SECONDARY OUTCOMES:
Improvement Rate of Glucose Metabolism in GDM Pregnant Women After Intervention | From participant enrollment (23-24+6 weeks of gestation) to 6 weeks postpartum
Long-term Incidence of Type 2 Diabetes Mellitus (T2DM) | From 6 months postpartum to 2 years postpartum
Incidence of Adverse Outcomes | From participant enrollment (23-24+6 weeks of gestation) to 6 weeks postpartum
Long-term Incidence of Cardiovascular Disease (CVD) | From 6 months postpartum to 2 years postpartum
Abnormal Blood Glucose Status in Offspring | From 6 months postpartum (6 months after offspring's birth) to 2 years postpartum (2 years after offspring's birth)
Obesity Rate in Offspring | From 6 months postpartum (6 months after offspring's birth) to 2 years postpartum (2 years after offspring's birth)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu women and children health hospital, Nanjing, China